CLINICAL TRIAL: NCT06592118
Title: Clinical Profiles, Surgical Strategies, and Outcomes of Follicular and Papillary Thyroid Carcinoma in Pediatric and Adolescent Populations: A Retrospective Comparative Study
Brief Title: Clinical and Surgical Outcomes of Thyroid Carcinoma in Children and Adolescents
Acronym: CPSO-TC
Status: Completed | Type: Observational
Sponsor: Dezhou Hospital Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: DZSRMYYZC2024095
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric and Adolescent Differentiated Thyroid Carcinoma; SEER Database Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FTC: Pediatric and Adolescent Patients with Follicular Thyroid Carcinoma
  Interventions: Other: Different Pathological Types (FTC vs PTC)
- PTC: Pediatric and Adolescent Patients with Papillary Thyroid Carcinoma
  Interventions: Other: Different Pathological Types (FTC vs PTC)

INTERVENTIONS:
Other: Different Pathological Types (FTC vs PTC) — Comprehensive Comparison of Pediatric and Adolescent Follicular Thyroid Carcinoma and Papillary Thyroid Carcinoma Patients
  Other Names: Different Pathological Types

SUMMARY:
This study aims to investigate the differences in clinical characteristics, causes of death, long-term survival, and surgical approaches between pediatric and adolescent follicular and papillary carcinoma by exploring data from the SEER database. The research is designed as a retrospective cohort study, primarily focused on collecting and comparing data to identify key disparities and outcomes between these two patient groups. It is anticipated that the findings will provide valuable insights into the management and prognosis of these cancers in younger populations, contributing to more targeted and effective treatment strategies.

DETAILED DESCRIPTION:
This study is a retrospective cohort analysis aimed at elucidating the differences between pediatric and adolescent patients diagnosed with follicular and [specific type] carcinoma, utilizing data sourced from the SEER (Surveillance, Epidemiology, and End Results) database. The focus of the research is on a comprehensive comparison of various clinical aspects, including demographic characteristics, tumor features, treatment modalities, and survival outcomes.

Key areas of investigation include the examination of clinical characteristics such as tumor size, location, and stage at diagnosis, as well as treatment approaches including surgery types and their impact on patient outcomes. Additionally, the study will assess the causes of death and overall survival rates among these young patients, aiming to identify any significant prognostic factors.

By leveraging the robust and extensive data available in the SEER database, this study seeks to uncover critical insights into the management of follicular and [specific type] carcinoma in pediatric and adolescent populations. The findings are expected to contribute to the development of more tailored and effective therapeutic strategies, ultimately improving long-term survival and quality of life for affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of Follicular Thyroid Carcinoma (FTC) or Papillary Thyroid Carcinoma (PTC).
* Age range: Pediatric and adolescent patients (ages 1-18 years).

Exclusion Criteria:

* Patients with incomplete survival and clinical information.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of pediatric and adolescent patients, aged 1 to 18 years, who have been diagnosed with Follicular Thyroid Carcinoma (FTC) or Papillary Thyroid Carcinoma (PTC). These patients were identified from a comprehensive database containing clinical, pathological, and surgical records.The population spans a diverse demographic, representing various ethnicities, genders, and geographical locations. This cohort was selected to ensure a thorough investigation of the differences in clinical presentations, surgical outcomes, and prognostic factors between the two types of thyroid carcinoma within the pediatric and adolescent age groups.
Sampling Method: Non-Probability Sample
Enrollment: 3068 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 20 years post-diagnosis
  Time from diagnosis until death from any cause.
T (Tumor) - Primary Tumor | Perioperatively/Periprocedurally
  T describes the size and/or extent of the primary tumor, T values typically range from T0 to T4, where T0 indicates no evidence of a primary tumor (not detectable), and T4 indicates a large tumor that has significantly invaded surrounding tissues.
N (Nodes) - Regional Lymph Nodes | Perioperatively/Periprocedurally
  The N staging will classify the extent of lymph node involvement as follows: N0 indicates no lymph node metastasis, N1a indicates metastasis to central compartment lymph nodes, and N1b indicates metastasis to lateral neck lymph nodes.
M (Metastasis) - Distant Metastasis | Within one month after the diagnosis of thyroid carcinoma
  M describes whether cancer has spread to other parts of the body (distant metastasis). M values are usually M0 or M1, where M0 indicates no distant metastasis, and M1 indicates the presence of distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Study Director — Qilu Hospital of Shandong University Dezhou

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) will be made available to other researchers under a formal data-sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication of the main study results and will be accessible for a period of 2 years.
Access Criteria: Researchers seeking access to the IPD must submit a methodologically sound proposal. Requests should be directed to the principal investigator and will be evaluated on the basis of scientific merit and ethical considerations.

REFERENCES:
- [Background] Cistaro A, Quartuccio N, Garganese MC, Villani MF, Altini C, Pizzoferro M, Piccardo A, Cabria M, Massollo M, Maghnie M, Campenni A, Siracusa M, Baldari S, Panareo S, Urso L, Bartolomei M, De Palma D, Grossi A, Mazzoletti A, Dondi F, Bertagna F, Giubbini R, Albano D. Prognostic factors in children and adolescents with differentiated thyroid carcinoma treated with total thyroidectomy and RAI: a real-life multicentric study. Eur J Nucl Med Mol Imaging. 2022 Mar;49(4):1374-1385. doi: 10.1007/s00259-021-05586-8. Epub 2021 Oct 19. PMID 34664092
- [Background] de Souza Reis R, Gatta G, de Camargo B. Thyroid carcinoma in children, adolescents, and young adults in Brazil: A report from 11 population-based cancer registries. PLoS One. 2020 May 1;15(5):e0232416. doi: 10.1371/journal.pone.0232416. eCollection 2020. PMID 32357198
- [Background] Moleti M, Aversa T, Crisafulli S, Trifiro G, Corica D, Pepe G, Cannavo L, Di Mauro M, Paola G, Fontana A, Calapai F, Cannavo S, Wasniewska M. Global incidence and prevalence of differentiated thyroid cancer in childhood: systematic review and meta-analysis. Front Endocrinol (Lausanne). 2023 Sep 19;14:1270518. doi: 10.3389/fendo.2023.1270518. eCollection 2023. PMID 37795368
- [Derived] Liu Y, Meng T, Ma S, Zheng Y, Miao Y, Zhang T. Clinical characteristics, surgical approaches, and prognosis of follicular and papillary thyroid cancer in children and adolescents: a retrospective cohort study. Pediatr Surg Int. 2025 Feb 28;41(1):89. doi: 10.1007/s00383-025-05990-3. PMID 40019558